CLINICAL TRIAL: NCT01275196
Title: ENESTChina: A Phase III Multi-center, Open-label, Randomized Study of Nilotinib Versus Imatinib in Chinese Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: Safety and Efficacy of Nilotinib vs. Imatinib in the Treatment of Newly Diagnosed Chinese Ph+ CML-CP Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ECN02
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Newly diagnosed,; Ph+ chronic myeloid leukemia,; CML-CP
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Imatinib Mesylate

ARMS (2):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib
- Imatinib (Active Comparator)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Nilotinib
  Arms: Nilotinib
Drug: Imatinib
  Arms: Imatinib

SUMMARY:
The study will compare the efficacy and safety of Nilotinib versus Imatinib in newly diagnosed Chinese patients with CML-CP.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chinese ethnicity greater than or equal to 18 years of age
* ECOG 0, 1, or 2.
* Patients with CML-CP (Ph+) within 6 months of diagnosis (date of initial diagnosis is the date of first cytogenetic analysis). Standard conventional cytogenetic analysis must be done on bone marrow. (FISH cannot be used)
* Diagnosis of chronic myelogenous leukemia in chronic phase with cytogenetic confirmation for the presence of Philadelphia chromosome of (9;22 translocation; less than 20 metaphases may be used for diagnosis
* Documented chronic phase CML will meet all the criteria defined by:

  * < 15% blasts in peripheral blood and bone marrow
  * < 30% blasts plus promyelocytes in peripheral blood and bone marrow
  * < 20% basophils in the peripheral blood
  * ≥ 100 x 109/L (≥ 100,000/mm3) platelets
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
* Adequate organ function as defined by:

  * Total bilirubin < 1.5 x ULN
  * SGOT and SGPT < 2.5 x ULN
  * Creatinine < 1.5 x ULN
  * Serum amylase and lipase ≤ 1.5 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related.
* Patients must have the following laboratory values (≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of study medication.):

  * Potassium ≥ LLN
  * Magnesium ≥ LLN
  * Phosphate ≥ LLN
  * Total calcium (corrected for serum albumin) ≥ LLN.
* Ability to provide written informed consent prior to any study related screening procedures being performed.

Exclusion Criteria:

* Patients with previously documented T315I mutations;
* Treatment with tyrosine kinase inhibitor(s) prior to study entry is not allowed, except in the following situation: in emergent cases where the patient requires disease management while awaiting study start, commercial supplies of Gleevec/Glivec at any dose may be prescribed to the patient but for no longer than 2 weeks in duration.
* Treatment with IFN for more than 3 months.
* Impaired cardiac function including any one of the following:
* Complete left bundle branch block
* Long QT syndrome or a known family history of long QT syndrome.
* History of or presence of clinically significant ventricular or atrial tachyarrhythmias
* Clinically significant resting bradycardia (<50 beats per minute)
* QTc > 450 msec If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
* History of clinically documented myocardial infarction within past 12 months
* History of unstable angina (during the last 12 months)
* Other clinically significant heart disease (e.g., congestive heart failure or uncontrolled hypertension).
* Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
* History of significant congenital or acquired bleeding disorder unrelated to cancer.
* Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery.
* Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 30 days of Day 1.
* History of non-compliance to medical regimens or inability to grant consent.
* Patients with another primary malignancy except if the other primary malignancy is neither currently clinically significant or requiring active intervention
* Patients actively receiving therapy with strong CYP3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. See link for complete list of these medications: http://medicine.iupui.edu/flockhart/table.htm or reference Protocol post text appendix 1.
* Patients actively receiving therapy with strong CYP3A4 inducers (e.g., dexamthasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbitol, St. John's Wort) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. See link for complete list of these medications: http://medicine.iupui.edu/flockhart/table.htm or reference Protocol post text appendix 1.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
* Acute or chronic liver, pancreatic or severe renal disease considered unrelated to disease.
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug (Please see http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm for a comprehensive list of agents that prolong the QT interval).
* Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) female of childbearing potential unwilling to use contraceptive precautions throughout the trial (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Fuzhou
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai

REFERENCES:
- [Derived] Wang J, Shen ZX, Saglio G, Jin J, Huang H, Hu Y, Du X, Li J, Meng F, Zhu H, Hu J, Wang J, Hou M, Hertle S, Menssen HD, Ortmann CE, Tribouley C, Yuan Y, Baccarani M, Huang X. Phase 3 study of nilotinib vs imatinib in Chinese patients with newly diagnosed chronic myeloid leukemia in chronic phase: ENESTchina. Blood. 2015 Apr 30;125(18):2771-8. doi: 10.1182/blood-2014-09-601674. Epub 2015 Mar 12. PMID 25766724

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized 1:1 between Nilotinib and Imatinib.
Groups:
- Imatinib: Patients received 400 mg qd (400 mg/day; may be increased to 600 mg/day).
- Nilotinib: Patients received 300 mg bid (600 mg/day)
Period: Overall Study
Arm/Group | Imatinib | Nilotinib
Started | 133 | 134
Intended to Continue Into Extension | 112 | 113
Completed | 113 | 113
Not Completed | 20 | 21
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Disease Progression | 6 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Suboptimal response/treatment failure | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib | Nilotinib | Total
Number analyzed (Participants) | 133 | 134 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (12.86) | 41.5 (12.76) | 40.6 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 43 | 95
  Male | 81 | 91 | 172

OUTCOME MEASURES:

1. Primary Outcome: Major Molecular Response (MMR) at 12 Months - With Imputation.
Description: Major molecular response (MMR) was defined as a value of ≤ 0.1% of BCR-ABL ratio on the IS. The minimum number of control genes for a sample to be valid was 3000. For statistical comparison purpose, MMR was considered as a binary variable with patients achieving MMR grouped as 'responders' and patients not achieving MMR, patients with missing PCR evaluations or patients with atypical transcripts at baseline grouped as 'non-responders'. This endpoint was calculated based on the 12 month analysis.
Time Frame: 12 months
Population: Patients in the FAS consisted of all patients who were randomized into the study. Following the intent-to-treat principle, patients were analyzed according to the treatment group to which they were assigned at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of Participants | 27.8 [20.4 to 36.3] | 52.2 [43.4 to 60.9]
Statistical Analysis 1: Comparison: Imatinib vs Nilotinib; Test type: Non-Inferiority or Equivalence — This trial was powered to detect an odds ratio of at least 2.333 which corresponds, for example, to increases of 18% (from 22% to 40%) and increases of 20% (from 30% to 50%); p = 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: MMR Rate at Each Time Point
Description: Major molecular response (MMR) was defined as a value of ≤ 0.1% of BCR-ABL ratio on the IS. The minimum number of control genes for a sample to be valid was 3000. For statistical comparison purpose, MMR was considered as a binary variable with patients achieving MMR grouped as 'responders' and patients not achieving MMR, patients with missing PCR evaluations or patients with atypical transcripts at baseline grouped as 'non-responders'. These time points including the 12 month data were calculated based on the final analysis after the end of the study.
Time Frame: Months 3,6,9,12,15, 18, 21, 24, 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of Participants
  3 Months | 3.0 [0.8 to 7.5] | 13.4 [8.2 to 20.4]
  6 Months | 18.0 [11.9 to 25.6] | 44.8 [36.2 to 53.6]
  9 Months | 21.1 [14.5 to 29.0] | 47.8 [39.1 to 56.6]
  12 Months | 27.8 [20.4 to 36.3] | 53.0 [44.2 to 61.7]
  15 Months | 36.1 [27.9 to 44.9] | 59.0 [50.1 to 67.4]
  18 Months | 40.6 [32.2 to 49.5] | 57.5 [48.6 to 66.0]
  21 Months | 41.4 [32.9 to 50.2] | 61.9 [53.2 to 70.2]
  24 Months | 49.6 [40.8 to 58.4] | 61.9 [53.2 to 70.2]
  36 Months | 59.4 [50.5 to 67.8] | 68.7 [60.1 to 76.4]

3. Secondary Outcome: Best MMR by Each Timepoint
Description: Best MMR rates by scheduled time point are cumulative response rates up to that time point. In this analysis, patients who had achieved MMR at or before the time point were counted as responders, no matter if they lost the response/discontinued or not. Therefore, this response rate represented the best observed response rate up to that specific time point.
Time Frame: Months 3,6,9,12,15, 18, 21, 24, 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of Participants
  Overall | 66.9 [58.2 to 74.8] | 73.9 [65.6 to 81.1]
  Month 3 | 3.0 [0.8 to 7.5] | 13.4 [8.2 to 20.4]
  Month 6 | 18.0 [11.9 to 25.6] | 45.5 [36.9 to 54.3]
  Month 9 | 22.6 [15.8 to 30.6] | 51.5 [42.7 to 60.2]
  Month 12 | 30.8 [23.1 to 39.4] | 56.0 [47.1 to 64.5]
  Month 15 | 37.6 [29.3 to 46.4] | 62.7 [53.9 to 70.9]
  Month 18 | 42.9 [34.3 to 51.7] | 64.2 [55.4 to 72.3]
  Month 21 | 46.6 [37.9 to 55.5] | 66.4 [57.8 to 74.3]
  Month 24 | 52.6 [43.8 to 61.3] | 67.9 [59.3 to 75.7]
  Month 36 | 65.4 [56.7 to 73.4] | 73.9 [65.6 to 81.1]

4. Secondary Outcome: Kaplan-Meier Estimates of Time to First MMR
Description: Time to first MMR (months) = (date of first MMR or censoring - date of randomization + 1) / 30.4375.
Time Frame: End of study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
months | 21.7 [16.5 to 25.2] | 8.1 [5.6 to 11.1]

5. Secondary Outcome: Durable MMR Rate at 24 Months
Description: The rate of durable MMR at 24 months, defined as the proportion of patients who have achieved MMR at 12 months, and also maintain continuous MMR until the 24 month time point (1 month = 28 days) without intervening loss of MMR in between 12 and 24 months
Time Frame: 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Perentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Perentage of Participants | 27.8 [20.4 to 36.3] | 50.7 [42.0 to 59.5]

6. Secondary Outcome: Kaplan-Meier Estimates of Duration of First MMR Among Patients Who Achieved MMR
Description: Duration of first MMR (months) = (date of loss of MMR or censoring-date of first MMR + 1)/30.4375.
Time Frame: End of Study (Up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.

7. Secondary Outcome: Best Complete Cytogenic Response (CCyR) Rate by Each Time Point
Description: CCyR is defined as 0% Ph+ metaphases based on at least 20 metaphases from bone marrow cytogenetics.
Time Frame: Months 6, 12, 18, 30, 24, 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of Participants
  Overall | 89.5 [83.0 to 94.1] | 85.8 [78.7 to 91.2]
  Month 6 | 57.1 [48.3 to 65.7] | 66.4 [57.8 to 74.3]
  Month 12 | 80.5 [72.7 to 86.8] | 77.6 [69.6 to 84.4]
  Month 18 | 84.2 [76.9 to 90.0] | 80.6 [72.9 to 86.9]
  Month 30 | 88.0 [81.2 to 93.0] | 84.3 [77.0 to 90.0]
  Month 24 | 86.5 [79.5 to 91.8] | 83.6 [76.2 to 89.4]
  Month 36 | 89.5 [83.0 to 94.1] | 85.8 [78.7 to 91.2]

8. Secondary Outcome: Kaplan-Meier Estimates of Time to First CCYR
Description: Time to first CCyR (months) = (date of first CCyR - date of randomization + 1) / 30.4375.
Time Frame: End of study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
months | 6.1 [5.6 to 6.6] | 5.6 [5.6 to 6.2]

9. Secondary Outcome: Kaplan-Meier Estimates of Duration of First CCyR Among Patients Who Achieved CCyR
Description: Duration of CCyR (months) = (date of CCyR loss or censoring-date of first CCyR + 1)/30.4375
Time Frame: End of Study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.

10. Secondary Outcome: Kaplan-Meier Estimates of Time to Progression to Accelerated Phase/Blast Crisis (AP/BC) on Treatment
Description: Time to progression to AP/BC was defined as the time from the date of randomization to the date of event defined as the first disease progression to AP/BC or the date of CML-related death, whichever is earlier. This variable was analyzed in 2 ways:
  * On-treatment: included progressions to AP/BC or CML-related deaths occurring on treatment in the study as events. The time was censored at the date of last on-treatment assessment (hematology, extramedullary disease, or cytogenetic evaluation) in the study for patients without event.
  * On-study: included progressions to AP/BC or CML-related deaths occurring in the study or during the follow-up period after discontinuation of treatment as events. The time was censored at the last assessment date in the study for patients who were still being treated and at the date of last contact for patients who discontinued treatment
Time Frame: End of study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.

11. Secondary Outcome: Kaplan-Meier Estimates of Event-free Survival (EFS) on Treatment
Description: Event-free survival was defined as the time from the date of randomization to the date of first occurrence of any of the following:-Death due to any cause, - Progression to AP or BC, Loss of partial cytogenetic response (PCyR), - Loss of CCyR, - Loss of CHR
Time Frame: End of Study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.

12. Secondary Outcome: Kaplan-Meier Estimates of Progression-free Survival (PFS) on Treatment
Description: Progression-free survival was defined as the time from the date of randomization to the date of event defined as the first disease progression to AP/BC or the date of death from any cause, whichever is earlier. This variable was analyzed in 2 ways:
  * On-treatment: included progressions to AP/BC or deaths occurring only on-treatment in the study as events. The time was censored at the date of last on-treatment assessment (hematology, extramedullary disease or cytogenetic evaluation) in the study before the cut-off date of the analysis for patients without event.
  * On-study: included progressions to AP/BC or deaths occurring in the study or during the follow-up period after discontinuation of study treatment as events. The time was censored at the last assessment date in the study for patients who were still being treated and at the date of last contact for patients who discontinued treatment.
Time Frame: End of study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — The median was not reached. | NA [NA to NA] — The median was not reached.

13. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival (OS) on Treatment
Description: Patients who discontinued study treatment early or completed the study protocol and did not enter into the extension protocol were to be followed for survival every 3 months for up to 2 calendar years from the date the last patient randomized received the first dose of study drug and every 6 months until Last Patient Last Visit. Overall survival (all deaths) was defined as the time between date of randomization and date of death due to any cause at any time during the study, including the follow-up period after discontinuation of treatment, i.e. overall survival on-study. The time was censored at the date of last assessment in the study for patients who are still being treated and at the date of last contact for patients who discontinued treatment.
Time Frame: End of Study (up to 40 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Months | NA [NA to NA] — Median could not be reached. | NA [NA to NA] — Median could not be reached.

14. Secondary Outcome: Best Complete Hematologic Response (CHR)
Description: CHR was defined as having all of the following criteria present at any assessment, which was confirmed by another assessment at least after 4 weeks: • WBC count < 10 x 10E9 /L • Platelet count < 450 x 10E9 /L • Basophils < 5% • No blasts and promyelocytes in peripheral blood • Myelocytes + metamyelocytes < 5 % in peripheral blood • No evidence of extramedullary involvement. The assessment was not considered CHR, if there were any values indicative of CML in AP or BC (i.e. by blasts in bone marrow). For confirmation of CHR, both the initial CHR as well as the confirming assessment (at least 4 weeks after the initial assessment) had to satisfy all criteria mentioned above, without any assessment in between which indicated 'No response'.
Time Frame: Months 1, 3, 4, 5, 6, 9,12, 15,18, 21, 24, 30, 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of participants
  Overall | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]
  Month 1 | 66.2 [57.5 to 74.1] | 73.1 [64.8 to 80.4]
  Month 3 | 91.0 [84.8 to 95.3] | 91.8 [85.8 to 95.8]
  Month 4 | 93.2 [87.5 to 96.9] | 93.3 [87.6 to 96.9]
  Month 5 | 94.0 [88.5 to 97.4] | 93.3 [87.6 to 96.9]
  Month 6 | 94.7 [89.5 to 97.9] | 93.3 [87.6 to 96.9]
  Month 9 | 94.7 [89.5 to 97.9] | 93.3 [87.6 to 96.9]
  Month 12 | 94.7 [89.5 to 97.9] | 94.0 [88.6 to 97.4]
  Month 15 | 94.7 [89.5 to 97.9] | 94.0 [88.6 to 97.4]
  Month 18 | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]
  Month 21 | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]
  Month 24 | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]
  Month 30 | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]
  Month 36 | 94.7 [89.5 to 97.9] | 94.8 [89.5 to 97.9]

15. Secondary Outcome: Modified ELN2009 Criteria
Description: Patients satisfying criteria for several "modified ELN 2009" categories are presented once under the worst category (Optimal> Suboptimal > Treatment failure). Patients in the "Discontinued" category are those who discontinued before the time point considered without satisfying any of the ELN 2009 criteria. Patients in the "Missing" category are those ongoing in the trial at the time point considered but with only missing or non evaluable data for ELN 2009 criteria.
Time Frame: End of Study (up to 40 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 133 | 134
Percentage of Participants
  Optimal Response | 39.8 | 55.2
  Suboptimal Response | 41.4 | 24.6
  Treatment Failure | 16.5 | 14.9
  Discontinued | 2.3 | 5.2

16. Secondary Outcome: Actual Dose Intensity
Description: Total dose/time on treatment (periods of zero dose were included).
Time Frame: End of Study (up to 40 months)
Population: Safety set consisted of all randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Imatinib | Nilotinib
Number analyzed (Participants) | 132 | 133
mg/day | 416.0 (62.40) | 536.4 (99.07)

17. Secondary Outcome: Summary Statistics of Trough Imatinib and Major Metabolite CGP74588 of Imatinib and Nilotinib PK Concentration by Time Point
Description: Pharmacokinetic Analysis Set
Time Frame: 12 Months
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CGP74588: Major metabolite of Imatinib
Arm/Group | Imatinib | CGP74588 | Nilotinib
Number analyzed (Participants) | 93 | 93 | 130
ng/mL
  Day 8 (Cycle 1) | 1235.3 (632.36) | 255.4 (154.74) | 1036.8 (618.10)
  Day 28 (Cycle 1) | 1291.3 (553.44) | 288.9 (130.25) | 970.4 (606.89)
  Day 84 (Cycle 3) | 1137.8 (461.50) | 235.7 (104.31) | 1172.4 (656.25)
  Day 168 (Cycle 6) | 1078.2 (413.99) | 243.2 (88.66) | 1154.8 (1034.15)
  Day 336 (Cycle 12) | 1111.1 (434.85) | 238.7 (89.11) | 1370.5 (878.88)
  Average trough PK | 1188.7 (452.24) | 258.7 (112.88) | 1137.4 (631.31)

ADVERSE EVENTS:
Description: The safety set consisted of all patients who received at least one dose of study medication. Two patients (1 in each arm) who were randomized but never treated were excluded from the safety set.
Groups:
- Imatinib 400 mg qd: Patients received 400 mg qd (400 mg/day; may be increased to 600 mg/day).
- Nilotinib 300 mg Bid: Patients received 300 mg bid (600 mg/day)
Arm/Group | Imatinib 400 mg qd | Nilotinib 300 mg Bid
Serious Adverse Events (participants affected / at risk) | 13/132 | 11/133
Other Adverse Events (participants affected / at risk) | 124/132 | 131/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400 mg qd (N=132) | Nilotinib 300 mg Bid (N=133)
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 3
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Blast cell count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Ovarian rupture (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400 mg qd (N=132) | Nilotinib 300 mg Bid (N=133)
Anaemia (Blood and lymphatic system disorders) | 18 | 12
Leukopenia (Blood and lymphatic system disorders) | 35 | 27
Neutropenia (Blood and lymphatic system disorders) | 18 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 37 | 41
Eyelid oedema (Eye disorders) | 25 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 18 | 5
Nausea (Gastrointestinal disorders) | 14 | 5
Vomiting (Gastrointestinal disorders) | 14 | 3
Face oedema (General disorders) | 11 | 0
Pyrexia (General disorders) | 15 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 40
Influenza (Infections and infestations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 25 | 17
Upper respiratory tract infection (Infections and infestations) | 13 | 10
Alanine aminotransferase increased (Investigations) | 16 | 28
Apolipoprotein B increased (Investigations) | 3 | 9
Aspartate aminotransferase increased (Investigations) | 9 | 13
Bilirubin conjugated increased (Investigations) | 3 | 15
Blood bilirubin increased (Investigations) | 8 | 41
Blood creatine phosphokinase increased (Investigations) | 12 | 6
Blood phosphorus decreased (Investigations) | 10 | 10
Gamma-glutamyltransferase increased (Investigations) | 3 | 15
Haemoglobin decreased (Investigations) | 14 | 8
Lipase increased (Investigations) | 29 | 37
Low density lipoprotein increased (Investigations) | 3 | 11
Neutrophil count decreased (Investigations) | 16 | 15
Platelet count decreased (Investigations) | 30 | 23
White blood cell count decreased (Investigations) | 28 | 16
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 16
Dizziness (Nervous system disorders) | 8 | 2
Headache (Nervous system disorders) | 4 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 17 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.